CLINICAL TRIAL: NCT02634034
Title: A Comparison Study to Evaluate the Pharmacokinetics and Safety of NK-104-CR in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kowa Research Institute, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: NK-104-CR-1.01US
Record Dates: First submitted 2015-12-10; First posted 2015-12-17 (Estimated); Last update posted 2016-01-11 (Estimated); Status verified 2016-01

CONDITIONS: Hyperlipidemia
MeSH Terms: conditions — Hyperlipidemias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- NK-104-CR (8mg), Pitavastatin IR (4mg), Pitavastatin IR (8mg) (Experimental)
  Interventions: Drug: A: NK-104-CR 8 mg; Drug: B: Pitavastatin IR 4 mg; Drug: C: Pitavastatin IR 8 mg
- Pitavastatin IR (4mg), Pitavastatin IR (8mg), NK-104-CR (8mg) (Experimental)
  Interventions: Drug: A: NK-104-CR 8 mg; Drug: B: Pitavastatin IR 4 mg; Drug: C: Pitavastatin IR 8 mg
- Pitavastatin IR (8mg), NK-104-CR (8mg), Pitavastatin IR (4mg) (Experimental)
  Interventions: Drug: A: NK-104-CR 8 mg; Drug: B: Pitavastatin IR 4 mg; Drug: C: Pitavastatin IR 8 mg

INTERVENTIONS:
Drug: A: NK-104-CR 8 mg — NK-104-CR 8 mg (Controlled Release single 8-mg tablet)
Drug: B: Pitavastatin IR 4 mg — Pitavastatin IR 4 mg (Immediate Release single 4-mg tablet)
Drug: C: Pitavastatin IR 8 mg — Pitavastatin IR 8 mg (Immediate Release two 4-mg tablets)

SUMMARY:
The purpose of this study is to compare the pharmacokinetics and safety of a controlled release (CR) version of pitavastatin (also referred to as NK-104) to immediate release (IR) pitavastatin in healthy adult volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Subject provides written informed consent before any study-specific evaluation is performed.
* Subject is a healthy adult male or female volunteer between the ages of 18 and 45 years, inclusive.
* Subject has no clinically significant abnormalities on the basis of medical history, physical examination findings, or vital sign measurements, as judged by the Investigator.
* Subject is able and willing to comply with the protocol and study procedures.

Exclusion Criteria:

* Subject is a woman who is pregnant or breastfeeding.
* Subject has clinically relevant abnormalities in the screening or check-in assessments.
* Subject has received an investigational drug within 30 days before the first dose of study drug.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2015-12; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Area Under the Curve | 0 to 48 hours
  Area Under the Curve 0 to tau

CONTACTS AND LOCATIONS:
Locations (1):
- Austin, Texas, United States